CLINICAL TRIAL: NCT03947944
Title: Clinical Outcomes of Small-incision Lenticule Extraction (SMILE) Using Vector Planning Method.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2018-0038
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Myopic Astigmatism
Keywords: Small incision lenticule extraction; astigmatism; vector planning
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manifest refraction planning group (Active Comparator): The subjects underwent SMILE using manifest refraction planning.
  Interventions: Procedure: SMILE using manifest refraction planning
- vector planning group (Active Comparator): The subjects underwent SMILE using vector planning.
  Interventions: Procedure: SMILE using vector planning

INTERVENTIONS:
Procedure: SMILE using manifest refraction planning — The treatments of astigmatism were planned using either the manifest refraction (manifest refraction group) or the vector planning method (vector planning group). The surgery was performed with standardized techniques with triple centration technique using the 500-KHz VisuMax system (Carl Zeiss Meditec AG, Jena, Germany). The superior cap depth was set as 120 µm, and the length of the side cut was set to 2 mm. Once the anterior (upper) and posterior (lower) planes of the lenticule were defined, the anterior and posterior interfaces were dissected using a microspatula with a blunt circular tip and extracted with microforceps. The integrity of the lenticule was assessed subsequently. The treatment plan for the vector planning group involved a combination of refractive astigmatism with 60 % emphasis and corneal astigmatism with 40 % emphasis.
  Arms: manifest refraction planning group
Procedure: SMILE using vector planning — The treatments of astigmatism were planned using either the manifest refraction (manifest refraction group) or the vector planning method (vector planning group). The surgery was performed with standardized techniques with triple centration technique using the 500-KHz VisuMax system (Carl Zeiss Meditec AG, Jena, Germany). The superior cap depth was set as 120 µm, and the length of the side cut was set to 2 mm. Once the anterior (upper) and posterior (lower) planes of the lenticule were defined, the anterior and posterior interfaces were dissected using a microspatula with a blunt circular tip and extracted with microforceps. The integrity of the lenticule was assessed subsequently. The treatment plan for the vector planning group involved a combination of refractive astigmatism with 60 % emphasis and corneal astigmatism with 40 % emphasis.
  Arms: vector planning group

SUMMARY:
In the past two decades, the femtosecond laser (FSL) technology has been introduced in the corneal refractive surgery filed, and brought a remarkable innovation. It can make tissue dissection through photodisruption and plasma cavitation. Initially, the FSL was used predominantly to make a corneal flap when performing laser in situ keratomileusis (LASIK), which is followed by stromal ablation using excimer laser. A new surgical technique called femtosecond lenticule extraction (FLEx) has been developed that uses only FSL to dissect two interfaces to create refractive lenticule and then remove it, which is very similar with LASIK. Small incision lenticule extraction (SMILE) which is the advanced form of all-in-one FSL refractive technique does not make a corneal flap rather make small incision where the separated refractive lenticule is removed through, and the upper part of the corneal tissue is called cap. Since the clinical outcomes of SMILE were firstly published in 2011, SMILE has been widely used for correction of myopia or myopic astigmatism worldwide. SMILE provides excellent visual outcomes and has advantages including a lesser decrease in corneal sensitivity and absence of flap related complications compared to LASIK.

The vector planning method is newly developed astigmatism correction method, which combines refraction astigmatism in 60 % emphasis and corneal astigmatism in 40 % emphasis. The vectorial difference between corneal astigmatism and refractive cylinder at the corneal plane is ocular residual astigmatism (ORA). In normal eyes treated for myopic astigmatism, the ORA typically ranges from 0.73 to 0.81 D. The eyes with high ORA resulted in inferior clinical outcomes after corneal refractive surgery including LASIK, LASEK, and SMILE. The vector planning method was effective in LASIK according to previous study. Therefore we try to confirm the efficacy of vector planning method in SMILE.

DETAILED DESCRIPTION:
Enrollment period : 6 months after IRB approval Participants : The subjects over 20 years old, who visited Severance hospital and Eyereum eye clinic for SMILE surgery with myopic astigmatism. The participants who satisfies criteria, and who can be monitored at all times during each period of observation after surgery are included in the study.

Methods: The subjects are randomly divided into two groups. One group underwent SMILE surgery using manifest refraction based planning, and the other group underwent SMILE surgery using vector planning. Before surgery, all patients underwent a detailed ophthalmological examination that included evaluation of logarithm of the minimum angle of resolution (logMAR) uncorrected-distance visual acuity (UDVA) and CDVA, manifest refraction, slit-lamp examination (Haag-Streit, Köniz, Switzerland), keratometry, and Scheimpflug-based corneal topography (Pentacam HR, Oculus). Dynamic corneal response (DCR) parameters were examined using Corvis ST. Corneal wavefront aberrations were measured using Keratron Scout (Optikon 2000, Rome, Italy). All examinations were repeated at 1, 3, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age of 20 years or older.
* 2. Myopia
* 3. Who is willing to get SMILE surgery

Exclusion Criteria:

* 1. Severe ocular surface disease
* 2. Any corneal disease, cataract, glaucoma, macular disease, or previous history of intraocular or corneal surgery
* 3. Patients with suspicion of keratoconus on corneal topography

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Uncorrected Distance Vision Acuity at each time point between the two groups. | preoperative
  Uncorrected Distance Vision Acuity in logMAR scale will be compared between the two groups at each time point.
Uncorrected Distance Vision Acuity at each time point between the two groups. | postoperative 6 months
  Uncorrected Distance Vision Acuity in logMAR scale will be compared between the two groups at each time point.
Corrected Distance vision Acuity at each time point between the two groups. | preoperative
  Corrected Distance Vision Acuity in logMAR scale will be compared between the two groups at each time point.
Corrected Distance vision Acuity at each time point between the two groups. | postoperative 6 months
  Corrected Distance Vision Acuity in logMAR scale will be compared between the two groups at each time point.

SECONDARY OUTCOMES:
Total higher order aberration at each time point between the two groups. | preoperative
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  1. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Total higher order aberration at each time point between the two groups. | postoperative 1 month
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  1. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Total higher order aberration at each time point between the two groups. | 3 months
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  1. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Total higher order aberration at each time point between the two groups. | 6 months
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  1. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Total higher order aberration changes from baseline at each postoperative time point between the two groups. | preoperative
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  2. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Total higher order aberration changes from baseline at each postoperative time point between the two groups. | postoperative 1 month
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  2. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Total higher order aberration changes from baseline at each postoperative time point between the two groups. | 3 months
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  2. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Total higher order aberration changes from baseline at each postoperative time point between the two groups. | 6 months
  Total higher order aberrations, spherical aberrations, and coma aberrations are examined using Keratron Scout (Optikon 2000, Rome, Italy). The unit of those is "μm".
  2. Total higher order aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Spherical aberration at each time point between the two groups. | preoperative
  3. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Spherical aberration at each time point between the two groups. | postoperative 1 month
  3. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Spherical aberration at each time point between the two groups. | 3 months
  3. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Spherical aberration at each time point between the two groups. | 6 months
  3. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Spherical aberration changes from baseline at each postoperative time point between the two groups. | preoperative
  4. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Spherical aberration changes from baseline at each postoperative time point between the two groups. | postoperative 1 month
  4. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Spherical aberration changes from baseline at each postoperative time point between the two groups. | 3 months
  4. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Spherical aberration changes from baseline at each postoperative time point between the two groups. | 6 months
  4. Spherical aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Coma aberration at each time point between the two groups. | preoperative
  5. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Coma aberration at each time point between the two groups. | postoperative 1 month
  5. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Coma aberration at each time point between the two groups. | 3 months
  5. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Coma aberration at each time point between the two groups. | 6 months
  5. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Coma aberration changes from baseline at each postoperative time point between the two groups. | preoperative
  6. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Coma aberration changes from baseline at each postoperative time point between the two groups. | postoperative 1 month
  6. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Coma aberration changes from baseline at each postoperative time point between the two groups. | 3 months
  6. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.
Coma aberration changes from baseline at each postoperative time point between the two groups. | 6 months
  6. Coma aberrations at each time point and change from baseline at each time point will be compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei Univeristy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No